CLINICAL TRIAL: NCT01467921
Title: A Randomized Phase II Study of Leucovorin, 5-fluorouracil With or Without Oxaliplatin (LV5FU2 vs. FOLFOX) for Curatively-resected, Node-positive Esophageal Squamous Cell Carcinoma.
Brief Title: Study of LV5FU2 Versus FOLFOX for Curatively-resected, Node-positive Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-07-206
Record Dates: First submitted 2011-11-06; First posted 2011-11-09 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Curatively-resected, Node-positive Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LV5FU2 (Active Comparator): leucovorin 200 mg/m2 and 5-fluorouracil 400 mg/m2 intravenously on day 1, followed by a 46-h protracted infusion of 5-fluorouracil 2,400 mg/m2
  Interventions: Drug: oxaliplatin
- FOLFOX (Experimental): leucovorin 200 mg/m2 and 5-fluorouracil 400 mg/m2 intravenously on day 1, followed by a 46-h protracted infusion of 5-fluorouracil 2,400 mg/m2 oxaliplatin 85 mg/m2 will be given intravenously on day 1 for over 2 h
  Interventions: Drug: oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin — oxaliplatin 85 mg/m2 will be given intravenously on day 1 for over 2 h

SUMMARY:
Oxaliplatin is a platinum analogue that has significant antitumor activity with better tolerability than cisplatin. The objective of the study is to evaluate the safety and activity of leucovorin and 5-fluorouracil and leucovorin and 5-fluorouracil plus oxaliplatin combination chemotherapy given as adjuvant therapy for curatively-resected, node-positive esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or older
* Histologically confirmed squamous cell carcinoma of esophagus
* Curatively (R0) resected, lymph node positive
* ECOG performance status of 0 or 1
* Restoration of oral intake >1500 kcal/d
* No prior chemotherapy except for neoadjuvant ones
* No prior radiotherapy within 1 month before registration
* Adequate marrow, hepatic, renal and cardiac functions
* Provision of a signed written informed consent

Exclusion Criteria:

* Severe co-morbid illness and/or active infections
* Prior treatment with oxaliplatin
* Pregnant or lactating women
* Active CNS metastases not controllable with radiotherapy or corticosteroids
* Known history of hypersensitivity to study drugs

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea